CLINICAL TRIAL: NCT04938037
Title: Comparison of Efficacy and Safety of Two Different Ultrasound-Guided Suprascapular Nerve Block Techniques in Chronic Shoulder Pain: A Prospective Double-Blinded Randomized Controlled Study
Brief Title: Comparison of the Efficacy of Two Different Suprascapular Nerve Block Techniques in Patients With Chronic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, İsa Cüce, Assistant professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/353
Record Dates: First submitted 2021-06-10; First posted 2021-06-24 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Chronic Shoulder Pain
Keywords: chronic shoulder pain; spinoglenoid notch; suprascapular nerve block; suprascapular notch
MeSH Terms: interventions — Methylprednisolone Acetate; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSNB through the spinoglenoid notch (Experimental): US guided 1ml methylprednisolone acetate (1ml / 40mg) and 5ml 0.5% bupivacaine Intervention: Medication: corticosteroids and local anesthetics
  Interventions: Procedure: US guided, SSNB with 1ml methylprednisolone acetate (1ml / 40mg) and 5 ml 0.5% bupivacaine
- SSNB through the suprascapular notch (Active Comparator): US guided 1ml methylprednisolone acetate (1ml / 40mg) and 5ml 0.5% bupivacaine Intervention: Medication: corticosteroids and local anesthetics
  Interventions: Procedure: US guided, SSNB with 1ml methylprednisolone acetate (1ml / 40mg) and 5 ml 0.5% bupivacaine

INTERVENTIONS:
Procedure: US guided, SSNB with 1ml methylprednisolone acetate (1ml / 40mg) and 5 ml 0.5% bupivacaine — nerve block

SUMMARY:
The aim of this study is to compare the efficacy and safety of the suprascapular nerve block (SSNB) at the spinoglenoid notch with SSNB at the suprascapular notch, which is the most commonly used technique in patients with chronic shoulder pain.

DETAILED DESCRIPTION:
Chronic shoulder pain (>3 months) is one of the most common musculoskeletal problems leading to psychosocial problems. Its causes include subacromial impingement, tendinosis, calcific tendinitis, complete or partial tendon tears, adhesive capsulitis, subacromial bursitis, glenohumeral osteoarthritis, glenohumeral instability, and acromioclavicular joint pathologies. For the treatment of chronic shoulder pain, conservative or surgical methods can be applied. Suprascapular nerve block (SSNB) is an effective and safe treatment option for pain relief and increases in functional activity in these patients.

The suprascapular nerve (SSN) is a peripheral nerve has both motor and sensory fibers, originates from the ventral rami of C5-C6 nerve roots. SSN passes across the posterior triangle of the neck and through the suprascapular notch enters to the supraspinous fossa. Then it comes to the infraspinous fossa via the spinoglenoid notch. The SSN has 3 sensory branches: a medial subacromial branch passes to the suprascapular notch, a lateral subacromial branch and a posterior glenohumeral branch pass the spinoglenoid notch. These branches supplies 70% of the sensory input to the shoulder.

In the literature, SSNB through suprascapular notch has positive effect on shoulder functions, pain and range of motion (ROM) in patients in the treatment of chronic shoulder pain. There is no study examining the efficacy of SSNB through spinoglenoid notch in the treatment of chronic shoulder pain.Therefore, the investigators planned this randomized trial to compare of the efficiency and safety of two different SSNB techniques (approach through suprascapular notch versus spinoglenoid notch) in treatment of patients with chronic shoulder pain.

Material and methods:

Participants: adult patients (>18 year old) with chronic shoulder pain Inclusion criteria: age ≥ 18 years old, shoulder pain that last more than 3 month, patients with a vas value of ≥ 4 despite treatment (drugs used for analgesia, local injections and physiotherapy methods), shoulder pain defined as non-specific shoulder pain, subacromial impingement syndrome, rotator cuff tendinopathy, adhesive capsulitis, non-traumatic instability, superior labrum anterior and posterior (SLAP) lesion, acromioclavicular pathology, shoulder osteoarthritis.

Exclusion criteria: A history of uncontrolled chronic diseases, e.g., malignant neoplasms, blood dyscrasia, previous surgery history at the affected shoulder, shoulder injection in the last 3 months before treatment, cervical radiculopathy or myelopathy, a previous fracture close to the shoulder region, septic arthritis or local infection in the affected shoulder, anaphylaxis against local anesthetics and/or corticosteroids, cardiac pacemaker, pregnancy.

Study Design: prospective, double blind, non-inferiority, randomized controlled trial Randomization method: 1:1 by computer randomization program

Detail of the intervention:

Experimental: SSNB through the spinoglenoid notch US guided 1ml methylprednisolone acetate (1ml / 40mg) and 5ml 0.5% bupivacaine Intervention: Medication: corticosteroids and local anesthetics Active comparator: SSNB through the suprascapular notch US guided 1ml methylprednisolone acetate (1ml / 40mg) and 5ml 0.5% bupivacaine Intervention: Medication: corticosteroids and local anesthetics

Outcome measurement:

Visual analogue scale of pain, active range of motion, shoulder pain and disability index (SPADI), Pain Pressure Threshold (PPT), Patient satisfaction

Statistical analyses:

Sample size calculation:

The sample size was calculated using http://statulator.com/SampleSize/ss2M.html considering a previous study. The non-inferiority margin for SPADI was taken as 9 points. Standard deviation 15.3 (assuming normal distribution) with a power of 80, an error of 0.05 type 1; 36 patients should be enrolled per groups. Including a rate of 10% drop-out 40 patients were planned to enroll in each groups.

Continuous variables

1. Student's t test: fit assumption of normal distribution
2. Mann-Whitney test: does not fit the assumption of normal distribution Categorical variables

1. Chi-square test 2. Fisher exact test: sparse data

The outcome differences within the experimental and active comparator groups of different time of evaluation will be analysed by using repeated-measures analysis of variance (ANOVA) with post hoc test with Bonferroni method.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Shoulder pain that last more than 3 month
3. Patients with a VAS value of ≥ 4 despite treatment (drugs used for analgesia, local injections and physiotherapy methods)
4. Shoulder pain defined as non-specific shoulder pain, subacromial impingement syndrome, rotator cuff tendinopathy, adhesive capsulitis, non-traumatic instability, SLAP lesion, acromioclavicular pathology, and / or shoulder osteoarthritis.

Exclusion Criteria:

1. A history of uncontrolled chronic diseases, e.g., malignant neoplasms, blood dyscrasia, and infection
2. Previous surgery history at the affected shoulder
3. Shoulder injection in the last 3 months before treatment
4. The presence of cervical radiculopathy or myelopathy
5. A previous fracture close to the shoulder region
6. Presence of septic arthritis or local infection in the affected shoulder
7. Presence of anaphylaxis against local anesthetics and / or corticosteroids
8. Presence of a cardiac pacemaker
9. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: İsa Cüce, Assist. Prof, Principal Investigator — Erciyes University Faculty of Medicine Hospital
Locations (1):
- Erciyes University Faculty of Medicine Hospital, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Background] Saglam G, Alisar DC. A Comparison of the Effectiveness of Ultrasound-Guided Versus Landmark-Guided Suprascapular Nerve Block in Chronic Shoulder Pain: A Prospective Randomized Study. Pain Physician. 2020 Nov;23(6):581-588. PMID 33185375
- [Background] Chan CW, Peng PW. Suprascapular nerve block: a narrative review. Reg Anesth Pain Med. 2011 Jul-Aug;36(4):358-73. doi: 10.1097/AAP.0b013e3182204ec0. PMID 21654552
- [Background] Laumonerie P, Blasco L, Tibbo ME, Bonnevialle N, Labrousse M, Chaynes P, Mansat P. Sensory innervation of the subacromial bursa by the distal suprascapular nerve: a new description of its anatomic distribution. J Shoulder Elbow Surg. 2019 Sep;28(9):1788-1794. doi: 10.1016/j.jse.2019.02.016. Epub 2019 Apr 26. PMID 31036420
- [Background] Vorster W, Lange CP, Briet RJ, Labuschagne BC, du Toit DF, Muller CJ, de Beer JF. The sensory branch distribution of the suprascapular nerve: an anatomic study. J Shoulder Elbow Surg. 2008 May-Jun;17(3):500-2. doi: 10.1016/j.jse.2007.10.008. Epub 2008 Feb 11. PMID 18262803
- [Background] Chang KV, Hung CY, Wu WT, Han DS, Yang RS, Lin CP. Comparison of the Effectiveness of Suprascapular Nerve Block With Physical Therapy, Placebo, and Intra-Articular Injection in Management of Chronic Shoulder Pain: A Meta-Analysis of Randomized Controlled Trials. Arch Phys Med Rehabil. 2016 Aug;97(8):1366-80. doi: 10.1016/j.apmr.2015.11.009. Epub 2015 Dec 14. PMID 26701762
- [Background] Shanahan EM, Ahern M, Smith M, Wetherall M, Bresnihan B, FitzGerald O. Suprascapular nerve block (using bupivacaine and methylprednisolone acetate) in chronic shoulder pain. Ann Rheum Dis. 2003 May;62(5):400-6. doi: 10.1136/ard.62.5.400. PMID 12695149

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SSNB Through the Spinoglenoid Notch | SSNB Through the Suprascapular Notch
Started | 40 | 40
Completed | 36 | 37
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SSNB Through the Spinoglenoid Notch | SSNB Through the Suprascapular Notch | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (9.3) | 57.2 (8.2) | 57.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 11 | 13 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 40 | 40 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI, kg/m2 [Mean (Standard Deviation); unit: Kg/m2] | 29.2 (5.6) | 30 (5.1) | 29.6 (5.3)
Affected shoulder, right [Count of Participants; unit: Participants] | 26 | 24 | 50
Symptom duration, months [Mean (Standard Deviation); unit: months] | 14.2 (9.5) | 15.6 (12.3) | 14.9 (11)

OUTCOME MEASURES:

1. Primary Outcome: Change of Shoulder Pain and Disability Index (SPADI)
Description: Shoulder pain and disability index (SPADI). The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability. Each item is scored between 0 and 10, and the resulting score is converted into a 100-point scale separately for pain, disability, and total score. Increased SPADI scores indicate an increase in patients' shoulder-related pain and disability.
Time Frame: Baseline and 1, 4, and 12 weeks after injection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SSNB Through the Spinoglenoid Notch | SSNB Through the Suprascapular Notch
Number analyzed (Participants) | 40 | 40
score on a scale
  SPADI- Total (Baseline- 1st week) | 22.1 (20.3) | 25.9 (23.7)
  SPADI- Total (Baseline- 4th week) | 27.0 (22.2) | 36.6 (22.0)
  SPADI- Total (Baseline- 12th week) | 29.4 (23.0) | 34.1 (28.1)
  SPADI - Pain (Baseline - 1st week) | 25.9 (22.2) | 27.5 (24.4)
  SPADI - Pain (Baseline - 4th week) | 29.4 (24.1) | 37.6 (21.7)
  SPADI - Pain (Baseline - 12th week) | 30.3 (26.0) | 35.7 (28.6)
  SPADI - Disability (Baseline - 1st week) | 20.3 (20.3) | 24.8 (24.5)
  SPADI - Disability (Baseline - 4th week) | 26.0 (22.3) | 35.8 (23.8)
  SPADI - Disability (Baseline - 12th week) | 29.6 (22.1) | 33.0 (29.2)

2. Secondary Outcome: Change of Visual Analog Scale (VAS)
Description: The degree of shoulder pain for night and activity was assessed using Visual Analog Scale (VAS) (range 0-10) for each patient. VAS was explained to the patients during assessment as 0 equal no pain and 10 equal worst imaginable pain.
Time Frame: Baseline and 1, 4, and 12 weeks after injection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SSNB Through the Spinoglenoid Notch | SSNB Through the Suprascapular Notch
Number analyzed (Participants) | 40 | 40
score on a scale
  VAS Activity (Baseline - 1st week) | 2.2 (2.5) | 2.8 (2.5)
  VAS Activity (Baseline - 4st week) | 2.8 (2.7) | 3.7 (2.4)
  VAS Activity (Baseline - 12th week) | 2.9 (2.7) | 3.5 (2.9)
  VAS Night (Baseline - 1st week) | 3.2 (2.6) | 3.0 (2.9)
  VAS Night (Baseline - 4st week) | 3.4 (2.6) | 3.9 (2.4)
  VAS Night (Baseline - 12th week) | 3.1 (2.7) | 3.3 (3.2)

3. Secondary Outcome: Change of Range of Motion (ROM)
Description: Active ROM of the affected shoulder is measured using a goniometer. These measurements included abduction, flexion, internal rotation, and external rotation.
Time Frame: Baseline and 1, 4, and 12 weeks after injection
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | SSNB Through the Spinoglenoid Notch | SSNB Through the Suprascapular Notch
Number analyzed (Participants) | 40 | 40
degree
  ROM flexion (Baseline- 1st week) | -3.9 (16.0) | -9.6 (14.0)
  ROM flexion (Baseline- 4th week) | -8.6 (18.3) | -18.6 (21.2)
  ROM flexion (Baseline- 12th week) | -8.8 (18.1) | -20.5 (22.2)
  ROM abduction (Baseline- 1st week) | -4.8 (14.4) | -9.6 (16.1)
  ROM abduction (Baseline- 4th week) | -14.1 (24.9) | -23.9 (30.1)
  ROM abduction (Baseline- 12th week) | -13.0 (27.7) | -26.0 (29.1)
  ROM internal rotation (Baseline- 1st week) | 0.9 (4.7) | -4.5 (9.7)
  ROM internal rotation (Baseline- 4th week) | -0.9 (3.2) | -7.5 (11.9)
  ROM internal rotation (Baseline- 12th week) | -2.4 (7.0) | -8.6 (12.2)
  ROM external rotation (Baseline- 1st week) | -2.5 (6.9) | -6.8 (17.3)
  ROM external rotation (Baseline- 4th week) | -6.0 (8.9) | -10.9 (16.0)
  ROM external rotation (Baseline- 12th week) | -8.5 (12.3) | -10.0 (20.3)

4. Secondary Outcome: Change of Pain Pressure Threshold (PPT)
Description: In order to determine the pain perception thresholds in the affected shoulder, Pain Pressure Threshold (PPT) values will be calculated by taking three measurements from the middle deltoid, upper trapezius, infraspinatus and tibialis anterior area with an algometer (Commander Echo® Algometer, JTECH Medical, Midvale, UT, USA). The average of the last 2 measurements will be taken and recorded. The PPT values were expressed as kilograms per square centimeter (kg/cm2). A low PPT value represents a decrease in the pain threshold and, therefore, increased sensitivity.
Time Frame: Baseline and 1, 4, and 12 weeks after injection
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | SSNB Through the Spinoglenoid Notch | SSNB Through the Suprascapular Notch
Number analyzed (Participants) | 40 | 40
kg/cm2
  PPT - upper trapezius (Baseline-1st week) | -0.3 (1.5) | 0.0 (1.5)
  PPT - upper trapezius (Baseline-4th week) | -0.1 (1.2) | -0.4 (1.4)
  PPT - upper trapezius (Baseline-12th week) | -0.2 (1.4) | -0.3 (1.3)
  PPT - middle deltoid (Baseline-1st week) | -0.2 (1.0) | 0.3 (1.5)
  PPT - middle deltoid (Baseline-4th week) | 0.0 (1.5) | 0.1 (1.8)
  PPT - middle deltoid (Baseline-12th week) | -0.2 (1.6) | -0.2 (1.6)
  PPT - Infraspinatus (Baseline-1st week) | -0.3 (1.4) | -0.1 (1.6)
  PPT - Infraspinatus (Baseline-4th week) | 0.0 (1.9) | -0.2 (1.6)
  PPT - Infraspinatus (Baseline-12th week) | -0.4 (1.7) | -0.2 (1.7)
  PPT - Tibialis Anterior (Baseline-1st week) | -0.3 (2.3) | -0.2 (1.4)
  PPT - Tibialis Anterior (Baseline-4th week) | -0.1 (1.9) | 0.1 (1.8)
  PPT - Tibialis Anterior (Baseline-12th week) | -0.4 (1.7) | -0.4 (1.5)

5. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction with the injection is determined by Likert Scale (1= very dissatisfied, 2= dissatisfied, 3=neither dissatisfied or satisfied, 4= satisfied, 5= very satisfied)
Time Frame: Assessed at baseline and 1, 4, and 12 weeks after injection, with week 12 reported.
Measure: Count of Participants; unit: Participants
Arm/Group | SSNB Through the Spinoglenoid Notch | SSNB Through the Suprascapular Notch
Number analyzed (Participants) | 40 | 40
Participants
  Extremely dissatisfied | 3 | 2
  Dissatisfied | 8 | 1
  neither dissatisfied or satisfied | 3 | 6
  Satisfied | 12 | 11
  Extremely satisfied | 14 | 20

ADVERSE EVENTS:
Time Frame: Adverse events up to the 12th week post-injection control were recorded.
Arm/Group | SSNB Through the Suprascapular Notch | SSNB Through the Spinoglenoid Notch
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 4/40 | 4/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSNB Through the Suprascapular Notch (N=40) | SSNB Through the Spinoglenoid Notch (N=40)
motor block (General disorders) | 1 (1) | 2 (2)
presyncope (General disorders) | 1 (1) | 1 (1)
redness and swelling at the injection site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
headache (General disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Chronic shoulder pain is a clinical spectrum that includes a heterogeneous group of diagnoses. The effectiveness of two different SSNB methods may differ in certain diagnostic groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT04938037/Prot_SAP_000.pdf